CLINICAL TRIAL: NCT05908955
Title: Efficacy and Safety of Quantitative Superior Vena Cava Isolation in Addition to Pulmonary Vein Isolation in Patients With Paroxysmal Atrial Fibrillation: the SCORE Randomized Controlled Trial
Brief Title: Quantitative Superior Vena Cava Isolation in Addition to Pulmonary Vein Isolation for Paroxysmal Atrial Fibrillation
Acronym: SCORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu,MD, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-GSP-GG-33
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: Radiofrequency ablation; Pulmonary vein; superior vena cava; clinical trial
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI (Active Comparator): Participants in this group will receive pulmonary vein isolation.
  Interventions: Procedure: PVI
- PVI+SVCI (Experimental): Participants in this group will receive superior vena cava isolation in addition to pulmonary vein isolation.
  Interventions: Procedure: PVI+ quantitative SVCI

INTERVENTIONS:
Procedure: PVI — pulmonary vein isolation
  Arms: PVI
Procedure: PVI+ quantitative SVCI — pulmonary vein isolation and superior vena cava isolation guided by quantitative ablation index
  Arms: PVI+SVCI

SUMMARY:
Pulmonary vein isolation (PVI) for paroxysmal atrial fibrillation (PAF) has limited success. The superior vena cava (SVC) has been identified as one of the most common non-pulmonary vein triggers for PAF. It is estimated that SVC isolation (SVCI) could improve the clinical results for patients with PAF. However, results from previous studies about SVCI remain controversial. It is possible that safety concerns for SVCI outweigh its benefits and lead to inadequate ablation. To address this issue, the introduction of a quantitative ablation index (AI) for SVCI may provide a solution.

The goal of this prospective, randomized controlled trial is to test the efficacy and safety of quantitative SVCI in addition to PVI in PAF. Participants with PAF will be randomly assigned to either PVI group or PVI+ quantitative SVCI group in a 1:1 ratio and will be followed up for 12 months. The main questions it aims to answer are:

1. Evaluate the efficacy of PVI+SVCI guided by quantitative AI.
2. Assess the safety of PVI+SVCI guided by quantitative AI.

The primary end point is treatment success at 3 months after the index ablation. The secondary end points include treatment success at 12 months, and safety outcomes.

DETAILED DESCRIPTION:
Catheter ablation has emerged as an effective treatment for drug-refractory PAF and is recommended as first-line therapy by current guidelines. PVI is considered the cornerstone of catheter ablation for atrial fibrillation (AF). However, despite persistent PVI, a subgroup of patients may experience recurrent AF due to focal ectopic discharges originating outside the pulmonary veins. Among the non-pulmonary vein triggers, the SVC stands out as a common culprit, making it a promising ablation target for maintaining sinus rhythm.

Nevertheless, results from previous studies that evaluate the efficacy of SVCI showed conflicting results. One possible explanation is that SVC is adjacent to critical anatomy structures (such as the sinus node and the phrenic nerve), which raises safety concerns and often leads to inadequate ablation.

Therefore, it is necessary to establish standardized ablation procedure for SVCI, ensuring both safety and efficacy. To address this issue, we proposed the concept of "quantitative ablation for SVCI." By introducing AI as a quantitative measure, it is possible to achieve precise catheter ablation while minimizing the risk of procedure-related complications.

The SCORE trial is single-center, prospective, randomized controlled trial aiming to enroll 290 patients with PAF. Participants with PAF will be randomly assigned to either PVI group or PVI+ quantitative SVCI group in a 1:1 ratio, and will be followed up for 12 months. The goal is to determine whether quantitative SVCI could improve clinical results for PAF when added to PVI. The key objectives are as follows:

1. Evaluate the efficacy of PVI+SVCI guided by quantitative AI.
2. Assess the safety of PVI+SVCI guided by quantitative AI.

The primary endpoint of the study is treatment success, defined as freedom from AF, atrial flutter, or atrial tachycardia lasting longer than 30 seconds, at the 3-month follow-up. Secondary endpoints include treatment success at the 12-month follow-up and safety outcomes, including death, stroke/TIA, pericardial tamponade or effusion requiring drainage, pulmonary vein stenosis, superior vena cava stenosis, diaphragmatic nerve injury or paralysis, sinus node dysfunction, and atrial esophageal fistula.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal AF that are unresponsive to antiarrhythmic drugs (one or more than one).
* Willing to undergo catheter ablation for AF.
* Age: 40-75 years old.

Exclusion Criteria:

* History of any type of catheter ablation for cardiac arrhythmias.
* History of any type of thoracic surgery, including cardiac surgery.
* History of malignant tumors.
* History of permanent pacemaker implantation.
* Peripherally inserted central catheter for long-term
* Heart failure (left ventricular ejection fraction ≤40% or NYHA class III~IV).
* Sinus node dysfunction
* Allergy to contrast agents.
* Pregnancy or lactation.
* Age: <40yrs or >75yrs.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-03-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with maintenance of sinus rhythm measured by 14-day Holter ECG at 3 months follow-up | 3 months
  The proportion of patients that are freedom from AF, atrial flutter, or atrial tachycardia for longer than 30 seconds measured by 14-day Holter ECG at 3 months after the index ablation.

SECONDARY OUTCOMES:
Proportion of patients with maintenance of sinus rhythm measured by 14-day Holter ECG at 12 months follow-up | 12 months
  The proportion of patients that are freedom from AF, atrial flutter, or atrial tachycardia for longer than 30 seconds measured by 14-day Holter ECG at 12 months after the index ablation.
Incidence of treatment emergent adverse events post ablation | 12 months
  Incidence of treatment emergent adverse events that include death, stroke/TIA, pericardial tamponade or effusion that requires drainage, pulmonary vein stenosis, superior vena cava stenosis, diaphragmatic nerve injury or paralysis, sinus node dysfunction, and atrial esophageal fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Science, Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Z, Hu D. An epidemiological study on the prevalence of atrial fibrillation in the Chinese population of mainland China. J Epidemiol. 2008;18(5):209-16. doi: 10.2188/jea.je2008021. Epub 2008 Sep 8. PMID 18776706
- [Background] Mark DB, Anstrom KJ, Sheng S, Piccini JP, Baloch KN, Monahan KH, Daniels MR, Bahnson TD, Poole JE, Rosenberg Y, Lee KL, Packer DL; CABANA Investigators. Effect of Catheter Ablation vs Medical Therapy on Quality of Life Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1275-1285. doi: 10.1001/jama.2019.0692. PMID 30874716
- [Background] Corrado A, Bonso A, Madalosso M, Rossillo A, Themistoclakis S, Di Biase L, Natale A, Raviele A. Impact of systematic isolation of superior vena cava in addition to pulmonary vein antrum isolation on the outcome of paroxysmal, persistent, and permanent atrial fibrillation ablation: results from a randomized study. J Cardiovasc Electrophysiol. 2010 Jan;21(1):1-5. doi: 10.1111/j.1540-8167.2009.01577.x. Epub 2009 Sep 1. PMID 19732237
- [Background] Miyazaki S, Takigawa M, Kusa S, Kuwahara T, Taniguchi H, Okubo K, Nakamura H, Hachiya H, Hirao K, Takahashi A, Iesaka Y. Role of arrhythmogenic superior vena cava on atrial fibrillation. J Cardiovasc Electrophysiol. 2014 Apr;25(4):380-386. doi: 10.1111/jce.12342. Epub 2014 Jan 6. PMID 24320606
- [Background] Santangeli P, Zado ES, Hutchinson MD, Riley MP, Lin D, Frankel DS, Supple GE, Garcia FC, Dixit S, Callans DJ, Marchlinski FE. Prevalence and distribution of focal triggers in persistent and long-standing persistent atrial fibrillation. Heart Rhythm. 2016 Feb;13(2):374-82. doi: 10.1016/j.hrthm.2015.10.023. Epub 2015 Oct 23. PMID 26477712
- [Background] Da Costa A, Levallois M, Romeyer-Bouchard C, Bisch L, Gate-Martinet A, Isaaz K. Remote-controlled magnetic pulmonary vein isolation combined with superior vena cava isolation for paroxysmal atrial fibrillation: a prospective randomized study. Arch Cardiovasc Dis. 2015 Mar;108(3):163-71. doi: 10.1016/j.acvd.2014.10.005. Epub 2015 Feb 7. PMID 25662699
- [Background] Ejima K, Kato K, Iwanami Y, Henmi R, Yagishita D, Manaka T, Fukushima K, Arai K, Ashihara K, Shoda M, Hagiwara N. Impact of an Empiric Isolation of the Superior Vena Cava in Addition to Circumferential Pulmonary Vein Isolation on the Outcome of Paroxysmal Atrial Fibrillation Ablation. Am J Cardiol. 2015 Dec 1;116(11):1711-6. doi: 10.1016/j.amjcard.2015.09.005. Epub 2015 Sep 10. PMID 26434513
- [Background] Sharma SP, Sangha RS, Dahal K, Krishnamoorthy P. The role of empiric superior vena cava isolation in atrial fibrillation: a systematic review and meta-analysis of randomized controlled trials. J Interv Card Electrophysiol. 2017 Jan;48(1):61-67. doi: 10.1007/s10840-016-0198-2. Epub 2016 Oct 14. PMID 27743289
- [Background] Higuchi K, Yamauchi Y, Hirao K, Marrouche NF. The importance of superior vena cava isolation in ablation strategy for atrial fibrillation. Curr Opin Cardiol. 2013 Jan;28(1):2-6. doi: 10.1097/HCO.0b013e32835b099b. PMID 23128496
- [Background] Zhang T, Wang Y, Liang Z, Zhao H, Han Z, Wang Y, Wu Y, Ren X. Effect of Combined Pulmonary Vein and Superior Vena Cava Isolation on the Outcome of Second Catheter Ablation for Paroxysmal Atrial Fibrillation. Am J Cardiol. 2020 Jun 15;125(12):1845-1850. doi: 10.1016/j.amjcard.2020.03.030. Epub 2020 Apr 3. PMID 32305224
- [Background] Yamashita S, Tokuda M, Isogai R, Tokutake K, Yokoyama K, Narui R, Kato M, Tanigawa S, Inada K, Matsuo S, Miyanaga S, Sugimoto K, Yoshimura M, Yamane T. Spiral activation of the superior vena cava: The utility of ultra-high-resolution mapping for caval isolation. Heart Rhythm. 2018 Feb;15(2):193-200. doi: 10.1016/j.hrthm.2017.09.035. Epub 2017 Sep 22. PMID 28943481
- [Background] Miyazaki S, Taniguchi H, Kusa S, Uchiyama T, Hirao K, Iesaka Y. Conduction recovery after electrical isolation of superior vena cava--prevalence and electrophysiological properties. Circ J. 2013;77(2):352-8. doi: 10.1253/circj.cj-12-0951. Epub 2012 Oct 23. PMID 23090663
- [Derived] Guan W, Li X, Chen K, Yao Y, Liu J. Anatomical variation of femoral vessels and ultrasound-guided femoral vein puncture for catheter ablation of arrhythmias. Pacing Clin Electrophysiol. 2024 Feb;47(2):330-335. doi: 10.1111/pace.14924. Epub 2024 Jan 19. PMID 38240379